CLINICAL TRIAL: NCT01140776
Title: OSNA Neoadjuvant Feasibility Study in Breast Cancer Patients
Brief Title: Clinical Evaluation of OSNA Breast Cancer System in Breast Cancer Patients Receiving Neoadjuvant Therapy
Status: Terminated | Type: Observational
Sponsor: Sysmex America, Inc. (Industry)
Responsible Party: Carrie Pineda, Sysmex America, Inc
Other Study IDs: OSNA-BC-NEO-001
Record Dates: First submitted 2010-06-03; First posted 2010-06-09 (Estimated); Last update posted 2011-06-07 (Estimated); Status verified 2011-06

CONDITIONS: Breast Neoplasms; Breast Diseases
Keywords: metastasis; molecular pathology
MeSH Terms: conditions — Breast Neoplasms; Breast Diseases; Neoplasm Metastasis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Samples of the tissue homogenate will be retained and may be used for for further testing.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- OSNA Breast Cancer System: For in vitro diagnostic use only.
  The OSNA Breast Cancer System is an automated semi-quantitative, in vitro diagnostic test for the rapid detection of greater than (>) 0.2 mm metastases in nodal tissue removed from sentinel lymph node biopsies of breast cancer patients. Results from the assay can be used to guide the intra-operative or post-operative decision to remove additional lymph nodes and to aid in patient staging. An assay positive + or ++ result indicates the presence of metastasis (> 0.2 mm). An assay positive ++ result predicts the presence of macrometastasis (> 2 mm).
  Post-operative histological evaluation of permanent sections of the tissue specimen, in accordance with usual diagnostic practice and using the Sysmex lymph node cutting scheme, is required.

SUMMARY:
The study will determine the sensitivity, specificity, negative predictive value and positive predictive value of the OSNA Breast Cancer System for patients receiving Sentinel Lymph Node biopsies after receiving neoadjuvant hormonal/chemotherapy as compared to permanent section Hematoxylin and Eosin (H&E) and Immuno-histochemistry (IHC) staining.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* 18 years of age or older
* Diagnosed pre-surgically with T1-T3 or T4 non-inflammatory breast cancer, clinically node positive or node negative upon clinical examination
* Scheduled for SLN biopsy after receiving neoadjuvant hormonal or chemotherapy
* Subjects (or the subjects' legal representatives) who have read, understood (to the best of their ability) and signed the informed consent form.

Exclusion Criteria:

* Pregnant subjects, confirmed by interview with either subject or treating physician
* Subjects previously diagnosed with other invasive cancer. Subjects with skin cancer (basal cell and squamous cell carcinoma) may be included, except for subjects diagnosed with melanoma
* Participation in other neoadjuvant protocols specifically requiring SLN biopsy prior to administration of neoadjuvant chemotherapy or hormonal therapy
* Subjects who have been judged to be an inappropriate candidate by any medical care provider (e.g., surgeon, oncologist or pathologist).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a previous diagnosis of breast cancer scheduled for sentinel lymph node dissection after receiving neoadjuvant hormonal/chemotherapy.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2010-11; Primary Completion 2012-07 (Estimated); Study Completion 2012-07 (Estimated)

PRIMARY OUTCOMES:
Prospectively assess the performance of the OSNA Breast Cancer System for the detection of SLN metastasis in subjects treated with neoadjuvant therapy prior to SLN biopsy by comparing results with standard histopathology evaluation. | 18 months

SECONDARY OUTCOMES:
Compare performance of the OSNA Breast Cancer System to intraoperative frozen section methods (mandatory) and imprint cytology methods (optional) with standard histopathology results from permanent sections. | 18 months
Correlate OSNA results and histology results with the status of non-sentinel lymph nodes. | 18 months
Determine incidence of breast cancer recurrence in axillary lymph nodes and distant organs within 5 years in study subjects (Phase II). | 18 months

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Arizona Cancer Center, Tucson, Arizona
  - University of Texas MD Anderson Cancer Center, Houston, Texas